CLINICAL TRIAL: NCT06503380
Title: Real-world Study on the Management of Hematological Toxicities Associated With Targeted Therapies for Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Other Study IDs: MA-CIM-RWS-001
Record Dates: First submitted 2024-06-18; First posted 2024-07-16 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Hematological Toxicity; Targeted Therapy; Breast Cancer
Keywords: Hematological toxicity; Targeted therapy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group: 1000 patients we are planning to observe will be included in one group.
  Interventions: Other: No intervenrion.

INTERVENTIONS:
Other: No intervenrion. — This study will respect the medication choices of researchers in the study, without specifying which medication to choose for treatment, dosage, mode of administration (including single drug, combination therapy, or sequential therapy), and duration of administration.

SUMMARY:
This multicenter, real-world, observational study will retrospectively and prospectively collect real-world data related to the investigational drugs. We plan to observe 1000 patients and collect data on treatment cycles N and N+1 of the targeted therapies. Retrospective data collection is based on existing patient diagnosis and treatment records, collecting information on patients who have completed two treatment cycles before January 1, 2024. Prospective data collection is based on routine clinical treatment during the study period, collected until the end of the next cycle of treatment or early termination of the study. To observe the disease characteristics and management mode of hematological toxicity related to targeted therapies of breast cancer, and explore the possible related factors of hematological toxicity, such as age, disease subtype, cancer stage, targeted therapy regimens, etc. This study will respect the medication choices of researchers in the study, without specifying which medication to choose for treatment, dosage, mode of administration (including single drug, combination therapy, or sequential therapy), and duration of administration.

ELIGIBILITY:
Inclusion Criteria:

* · The patients signed the informed consent and voluntarily participated in the study.

  * A definite diagnosis of any type of breast cancer.
  * Receiving or has completed targeted therapies.
  * Investigator judged that the patient need to receive or had received treatment or prevention for CTIT, CIN or CRA induced by targeted therapies.

Exclusion Criteria:

* · Pregnant or lactating women.

  * Failure to understand the study or to obtain informed consent.
  * The investigator determined other situations that are not suitable for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We plan to observe 1000 patients and collect data on treatment cycles N and N+1 of the targeted therapies. Retrospective data collection is based on existing patient diagnosis and treatment records, collecting information on patients who have completed two treatment cycles before January 1, 2024. Prospective data collection is based on routine clinical treatment during the study period, collected until the end of the next cycle of treatment or early termination of the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of cancer treatment induced neutropenia (CIN) | Approximately 2 years
  The occurrence, prevention, treatment of neutropenia associated with targeted therapies. The influence of different baseline characteristics of patients on treatment outcomes and efficacy and safety of drugs.

SECONDARY OUTCOMES:
Incidence of cancer therapy induced thrombocytopenia (CTIT) | Approximately 2 years
  Characteristics and management of thrombocytopenia induced by targeted therapies of breast cancer.
Incidence of cancer related anemia (CRA) | Approximately 2 years
  Characteristics and management of anemia induced by targeted therapies in breast cancer patients in the real world.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ming Shao, Principal Investigator — Fudan University
Locations (1):
- Zhi-Ming Shao, Shanghai, Not US/Canada, China